CLINICAL TRIAL: NCT05174572
Title: Index of Microcirculatory Resistance Evaluation in Patients with Coronary Sinus Reducer Implantation for the Treatment of Chronic Refractory Angina Pectoris, the INROAD Study
Brief Title: IMR Evaluation in Patients with Coronary Sinus Reducer Implantation (INROAD Study)
Acronym: INROAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Futuro in Ricerca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021
Record Dates: First submitted 2021-12-03; First posted 2021-12-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Refractory Angina Pectoris
Keywords: Angina; Microcirculation resistance; Coronary sinus Reducer
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMR (Other): IMR evaluation before and after Reducer implantation
  Interventions: Procedure: IMR

INTERVENTIONS:
Procedure: IMR — Patients undergoing coronary sinus reducer implantation (Reducer) undergo evaluation of the index of microcirculatory resistance (IMR) at the time of implantation, and at 4 months follow-up.

SUMMARY:
The INROAD is an investigator-driven, prospective, study in which patients undergoing coronary sinus reducer implantation (Reducer) for chronic refractory angina undergo evaluation of the index of microcirculatory resistance (IMR) at the time of implantation, and at 4 months follow-up

DETAILED DESCRIPTION:
Refractory angina (RA) is a chronic condition (present for at least 3 months) of moderate-severe symptoms (Canadian class Cardiovascular Society [CCS] II-IV) due to coronary artery disease which cannot be adequately controlled by the combination of optimal medical therapy and coronary revascularization. The clinical impact in terms of quality of life, re-hospitalization and socio-health costs is extremely negative. In this context, the therapeutic goals are primarily the management of the symptom and improvement the patient's quality of life. The unpaid therapeutic demand of these patients has brought out a large number of medical and interventional treatments, including the coronary sinus reduction system (REDUCER). Numerous clinical studies and registries have been carried out and they proved both the efficacy and safety in the use of REDUCER. The physiological mechanism that are supposed to be behind the antianginal effect of coronary sinus intervention are essentially two:

1. Redistribution of coronary flow from the subepicardium to the subendocardium.
2. Coronary neoangiogenesis In both cases, the primum movens of the Reducer's therapeutic mechanism is attributable to the increase in venous pressure due to narrowing of the coronary sinus. Nevertheless, this mechanism of action is theoretical and has never been objectively tested. The evaluation of microcirculatory resistance by IMR before and after REDUCER implantation could be the most effective way to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Chronic refractory angina refractory to medical and interventional therapies.
* At least one open coronary artery (excluded right coronary artery) where to performs IMR evaluation
* Ability to provide informed written consent
* Life expectancy ≥1 year

Exclusion Criteria:

* Recent (within 3 months) acute coronary syndrome
* Left ventricular ejection fraction of <30%
* Severe valvular heart disease
* Inability to perform IMR
* Technical contraindications to the implant ( A pacemaker electrode in the coronary sinus, Mean right atrial pressure >15mmHg, Anomalous coronary sinus anatomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in IMR value | 4 month after Reducer implantation
  Significant Change (≥ 20%) in index of microcirculatory resistance (IMR) value at 4 month follow-up as compared to baseline value (before Reducer implantation). The IMR is calculated by multiplying the distal coronary pressure by the mean transit time of a 3 ml bolus of saline at room temperature during coronary hyperaemia induced by intravenous adenosine. Normal values are usually reported as ≤25.

SECONDARY OUTCOMES:
Change in angina severity according to the Seattle Angina Questionnaire | 4 month after Reducer implantation
  Change in angina severity according to the Seattle Angina Questionnaire (SAQ) after Reducer implantation. The questionnaire is performed before the Reducer implantation and after 4 months. The scores on the SAQ angina frequency scale of 0-30 points indicate daily angina, 31-60 points indicate weekly angina, 61-99 points indicate monthly angina, and 100 points indicate no angina. Zero at SAQ indicate a worst clinical situation.
Change in Canadian Cardiovascular Society angina class a | 4 month after Reducer implantation
  Change in Canadian Cardiovascular Society (CCS) angina class by two or more classes after Reducer implantation. The CCS evaluation is performed before the Reducer implantation and after 4 months. A CCS angina class I: ordinary activity such as walking or climbing stairs does not precipitate angina. CCS II : angina precipitated by emnotion, cold weather or meals and by walking up stairs-. CCS III: marked limitation of ordinary physical activity. CCS III indicate a worst clinical situation.
Change in Beck depression inventory | 4 month after Reducer implantation
  Change in Beck depression inventory (BDI) scale after Reducer Implantation. The questionnaire is performed before the Reducer implantation and after 4 months. A BDI scores from 0 through 9 indicate no or minimal depression; scores from 10 through 18 indicate mild to moderate depression; scores from 19 through 29 indicate moderate to severe depression; and scores from 30 through 63 indicate severe depression.A BDI of 63 indicate a worst clinical situation.
Change in CFR (coronary flow reserve) | 4 month after Reducer implantation
  Change in CFR (coronary flow reserve) value after Reducer Implantation. The CFR is performed before the Reducer implantation and after 4 month. CFR is defined as hyperemic coronary flow divided by resting flow and can be measured invasively in the catheterization laboratory with a cut-off of normality ≥ 2.0.
Change in RRR (resistive reserve ratio) value | 4 month after Reducer implantation
  Change in RRR (resistive reserve ratio) value after Reducer implantation. The RRR is performed before Reducer implantation and after 4 month. RRR was calculated as the ratio between resting and hyperemic distal coronary pressure ([resting Tmn/hyperemic Tmn] × [resting Pd/ hyperemic Pd]); which can therefore be simplified as the relationship between CFR x [resting Pd/ hyperemic Pd]. Cut-off values of normality is > 3.5.
Change in LVEDP (left ventricular end-diastolic pressure) | 4 month after Reducer implantation
  Change in LVEDP (left ventricular end-diastolic pressure) after Reducer implantation. LVEDP is performed before Reducer implantation and after 4 month. The LVEDP is measure 50 ms after the beginning of the QRS complex, usually coinciding with the R wave. The normal LVEDP cut-off is 15 mmHg.
Change in Speckle tracking echocardiography (STE) value | 4 month after Reducer implantation
  Change in Speckle tracking echocardiography (STE) value after Reducer implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tebaldi M, Campo G, Ugo F, Guarracini S, Marrone A, Clo S, Abdirashid M, Di Mauro M, Rametta F, Di Marco M, Cocco M, Marchini F, Penzo C, Erriquez A, Banai S, Biscaglia S. Coronary Sinus Narrowing Improves Coronary Microcirculation Function in Patients With Refractory Angina: A Multicenter Prospective INROAD Study. Circ Cardiovasc Interv. 2024 Jan;17(1):e013481. doi: 10.1161/CIRCINTERVENTIONS.123.013481. Epub 2024 Jan 16. PMID 38227697